CLINICAL TRIAL: NCT01370863
Title: An Explorative, Randomized, Placebo-controlled, DB, Parallel-group Trial, to Evaluate the Pharmacodynamic Effect of SPD557 on Reflux Parameters in Subjects With GERD & With Persistent Symptoms Despite Taking a Stable Dose of PPIs
Brief Title: An Explorative Trial to Evaluate the Pharmacodynamic Effect of SPD557 on Reflux Parameters in Refractory GERD Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated early due to recruitment difficulties. There were no safety concerns.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPD557-202; 2010-021397-12 (EudraCT Number)
Record Dates: First submitted 2011-05-31; First posted 2011-06-10 (Estimated); Results first posted 2013-06-07 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; Gastroesophageal reflux disease; SPD557; Proton pump inhibitors
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPD557 (Experimental)
  Interventions: Drug: SPD557
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SPD557 — 0.5 mg tablet t.i.d. for 4 weeks on top of stable PPI treatment
  Arms: SPD557
Drug: placebo — matching placebo tablet t.i.d. for 4 weeks on top of stable PPI treatment
  Arms: Placebo

SUMMARY:
The purpose of this trial is to investigate the pharmacodynamic effect on reflux parameters of SPD557 tablets (0.5 mg t.i.d., on top of PPI treatment) in patients with Gastroesophageal Reflux Disease (GERD) with persistent symptoms despite taking a stable dose of proton pump inhibitors. Additionally the effect on symptoms will be explored and safety and tolerability will be evaluated.

ELIGIBILITY:
Inclusion criteria:

1. Written ICF signed voluntarily before the first trial related activity.
2. Subjects with a history of GERD symptoms (i.e., heartburn and/or regurgitation) during the last 6 months
3. Subjects on a stable dose of PPIs, compliant for at least 6 weeks prior to screening.
4. ≥3 days per week with heartburn and/or regurgitation symptoms of at least moderate severity and a minimum of 25 liquid containing reflux events over 24h (pH/MII monitoring).

Exclusion criteria:

1. Subjects with prior endoscopic anti-reflux procedure or major GI surgery or subjects with major GI disorders.
2. Presence of severe and clinically uncontrolled cardiovascular, liver or lung disease, neurologic, cancer or AIDS.
3. Alarm symptoms suggestive of malignancies or organic disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2010-12-02 (Actual); Primary Completion 2012-05-29 (Actual); Study Completion 2012-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (15):
- Belgium (3):
  - CUB Hôpital Erasme, Brussels, Brussels Capital
  - Cliniques universitaires Saint Luc, Brussels
  - UZ Leuven, Belgium, Leuven
- France (3):
  - CHU de Bordeaux - Hôpital Saint André, Bordeaux
  - CHU de Lyon - Groupement Hospitalier Edouard Herriot, Lyon
  - Hôtel Dieu - CHU de Nantes, Nantes
- Germany (2):
  - Klinikum Garmisch-Partenkirchen GmbH, Garmisch-Partenkirchen
  - Otto-von-Guericke University, Magdeburg
- Academisch Medisch Centrum (AMC), Amsterdam, Netherlands
- Switzerland (3):
  - Inselspital Bern (Bern University Hopsital), Bern
  - Kantonsspital St. Gallen, Sankt Gallen
  - University Hospital Zurich, Zurich
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge
  - Wingate Institute of Neurogastroenterology, London
  - Queen's Medical Center (Nottingham University Hospital), Nottingham

REFERENCES:
- [Derived] Tack J, Zerbib F, Blondeau K, des Varannes SB, Piessevaux H, Borovicka J, Mion F, Fox M, Bredenoord AJ, Louis H, Dedrie S, Hoppenbrouwers M, Meulemans A, Rykx A, Thielemans L, Ruth M. Randomized clinical trial: effect of the 5-HT4 receptor agonist revexepride on reflux parameters in patients with persistent reflux symptoms despite PPI treatment. Neurogastroenterol Motil. 2015 Feb;27(2):258-68. doi: 10.1111/nmo.12484. Epub 2014 Dec 21. PMID 25530111

RESULTS

PARTICIPANT FLOW:
Groups:
- SPD557: 0.5 mg tablet administered 3 times daily (t.i.d.) for 4 weeks in addition to stable proton pump inhibitor (PPI) treatment
- Placebo: Matching placebo tablet administered three times daily (t.i.d.) for 4 weeks in addition to stable PPI treatment
Period: Overall Study
Arm/Group | SPD557 | Placebo
Started | 34 | 33
Completed | 32 | 30
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Did not want second pH/MII monitoring | 1 | 1
Not completed — Not meeting inclusion/exclusion criteria | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population was used defined as all subjects randomized into the study with at least 1 administration of the investigational product. Two subjects never received investigational product (n = 65).
Groups:
- SPD557: 0.5 mg tablet t.i.d. for 4 weeks in addition to stable proton pump inhibitor (PPI) treatment
- Placebo: Matching placebo tablet t.i.d. for 4 weeks in addition to stable PPI treatment
- Total: Total of all reporting groups
Arm/Group | SPD557 | Placebo | Total
Number analyzed (Participants) | 34 | 31 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (16.04) | 45.8 (14.50) | 44.8 (15.24)
Age, Customized [Count of Participants; unit: Participants]
  Between 18 and 70 years inclusive | 34 | 31 | 65
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 15 | 14 | 29
Region of Enrollment [Count of Participants; unit: Participants] — All randomized subjects (n = 67).
  Participants
    France | 13 | 13 | 26
    Belgium | 8 | 7 | 15
    Netherlands | 2 | 3 | 5
    Germany | 4 | 4 | 8
    United Kingdom | 3 | 4 | 7
    Switzerland | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Number of Liquid-containing Reflux Events (pH/MII Monitoring) at 4 Weeks
Description: This is used to characterize gastric reflux events. The measurements were made over a 24-hour period at baseline and again at week 4.
Time Frame: Baseline and 4 weeks
Population: Pharmacodynamics Population (PD) defined as all randomized subjects with at least 1 administration of the investigational product and with both a baseline and post-baseline PD assessment.
Measure: Mean (Standard Deviation); unit: Number of Reflux Events
Arm/Group | SPD557 | Placebo
Number analyzed (Participants) | 31 | 29
Number of Reflux Events | -17.9 (59.88) | -13.7 (37.58)
Statistical Analysis 1: Comparison: SPD557 vs Placebo; Test type: Superiority or Other; p = 0.869, ANCOVA; Difference in LS Mean = -1.452, 95% CI 2-sided [-19.054 to 16.149]

2. Secondary Outcome: Change From Baseline in the Number of Days With Heartburn and/or Regurgitation at 4 Weeks
Time Frame: Baseline and 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | SPD557 | Placebo
Number analyzed (Participants) | 31 | 29
Number of days | -0.90 (1.434) | -0.88 (1.610)
Statistical Analysis 1: Comparison: SPD557 vs Placebo; Test type: Superiority or Other; p = 0.487, ANCOVA; Diference in LS means = 0.264, 95% CI 2-sided [-0.495 to 1.024]

3. Secondary Outcome: Change From Baseline in the Patient Assessment of Upper Gastrointestinal Symptom Severity Index (PAGI-SYM) Questionnaire at 4 Weeks
Description: The PAGI-SYM contains 20 items and the scores range from 0 (no symptoms)-5 (very severe symptoms) for each item with a total score of 0-100. Higher scores indicate more severe gastrointestinal symptoms.
Time Frame: Baseline and 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD557 | Placebo
Number analyzed (Participants) | 31 | 29
Units on a scale | -0.41 (0.943) | -0.37 (0.760)
Statistical Analysis 1: Comparison: SPD557 vs Placebo; Test type: Superiority or Other; p = 0.637, ANCOVA; Difference in LS means = -0.087, 95% CI 2-sided [-0.501 to 0.326]

ADVERSE EVENTS:
Description: The Safety Population was defined as all subjects randomized into the study with at least 1 administration of the investigational product. Two subjects never received investigational product (n = 65).
Arm/Group | SPD557 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/31
Other Adverse Events (participants affected / at risk) | 25/34 | 16/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPD557 (N=34) | Placebo (N=31)
Diarrhea (Gastrointestinal disorders) | 13 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Headache (Nervous system disorders) | 12 | 4
Dizziness (Nervous system disorders) | 2 | 2
Influenza (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 3 | 1
Pharyngitis (Infections and infestations) | 0 | 2
Edema peripheral (General disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
Results data should be interpreted with caution since the study's early termination affects the statistical power to detect true differences between treatment groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.